CLINICAL TRIAL: NCT05548231
Title: A Multiple Dose Escalation Study in Chinese Participants With Overweight BMI or Obesity to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3437943
Brief Title: A Study of LY3437943 in Chinese Participants With Obesity Or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17954; J1I-MC-GZBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY3437943 (Experimental): LY3437943 administered subcutaneously (SC)
  Interventions: Drug: LY3437943
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: LY3437943
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn about the safety and tolerability of LY3437943 when given to Chinese participants with overweight body mass index (BMI) or obesity. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Each enrolled participant will receive injections of LY3437943 or placebo given just under the skin. For each participant, the study will last about 20 weeks excluding screening period and may include up to 20 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

For All Participants:

* Are native Chinese males or females
* Have a body mass index of ≥27 and ≤40 kilograms per square meter (kg/m²)
* Have not modified diet or adopted any nutritional lifestyle modification for 3 months
* Have stable body weight for the last three months
* Male participants must agree to use contraception during the study and for 4 months afterward and female participants must be woman of nonchildbearing potential

For Type 2 Diabetes Mellitus (T2DM) Participants:

* Have type 2 diabetes for at least 3 months
* Have a glycated hemoglobin (HbA1c) value of ≥7.0% and ≤10.5% and have been treated with diet and exercise alone or a stable dose of metformin for at least 3 months prior to screening

Exclusion Criteria:

For All Participants:

* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week and smoke more than 10 cigarettes, or cigarette equivalent (as determined by investigator), per day
* Have other serious or unstable illnesses
* Have had an episode of severe hypoglycemia
* Current or chronic history of liver disease.

For T2DM Participants:

* Have type 1 diabetes mellitus
* Have uncontrolled diabetes, defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization
* Any glucose-lowering medications other than metformin within 3 months prior to screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 20
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3437943 | Predose through Day 109
  PK: Cmax of LY3437943
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3437943 | Predose through Day 109
  PK: AUC of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No